CLINICAL TRIAL: NCT02763371
Title: Cognition Intervention Study Dortmund- Glycemic Index (CogniDo GI)
Acronym: CogniDo-GI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: COG0416DO
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Cognitive Function
Keywords: high GI lunch; low GI lunch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary: high GI lunch (Experimental): High GI-rice lunch ad libitum on test day 1 and low GI-rice lunch on test day 2. Water at libitum was constantly available on both days.
  Interventions: Other: Dietary: high GI lunch
- Dietary: low GI lunch (Experimental): Low GI-rice lunch ad libitum on test day 1 and high GI-rice lunch on test day 2. Water at libitum was constantly available on both days.
  Interventions: Other: Dietary: low GI lunch

INTERVENTIONS:
Other: Dietary: high GI lunch — High GI: High-GI rice lunch ad libitum on test day 1 and low GI-rice lunch on test day 2. Water at libitum was constantly available on both days.
  Arms: Dietary: high GI lunch
Other: Dietary: low GI lunch — Low-GI: Low GI-rice lunch ad libitum on test day 1 and high GI-rice lunch on test day 2. Water at libitum was constantly available on both days.
  Arms: Dietary: low GI lunch

SUMMARY:
The Cognition Intervention Study Dortmund (CogniDo) and the Cognition Intervention Study Dortmund PLUS (CogniDo PLUS) investigated the short-term effects of having school lunch versus skipping it on children's basal (CogniDo) and executive (CogniDo PLUS) cognitive functions in the afternoon. The The Cognition Intervention Study Dortmund Continued (Coco) connected this two previous studies and investigates the effect of having school lunch versus skipping it on children's basal and executive cognitive functions later in the afternoon. The present study the Cognition Intervention Study Dortmund- Glycemic Index (CogniDo GI) examines the influence of the gylcemic index of lunch on cognitive performance of school children in the afternoon.

DETAILED DESCRIPTION:
Glucose is the main fuel of the human brain. However, which impact the glycemic index of lunch has on cognitive performance is not clear. A recently published review by Philippou and Constantinou suggested cautiously that a low-GI meal may favor cognitive functions in adults, but note that their findings are inconclusive due to differences in study design, study sample (e.g. size, age), time of testing and the cognitive domain being examined. Because of cerebral particularities, children may react highly sensitive to variations of glycose supply. Therefore, an optimised composition of meals at favourable mealtime should be considered for optimal cognitive performance. The increasing implementation of all-day schools in Germany requires the children's catering for lunch at school.

As prior intake of food can have an influence on the physiological effect of test meal, the children's dietary intake in the mid-morning is standardized. The intervention is integrated in everyday school life: 9.15 a.m. standardized snack within the frame of the regular break, 9.45 a.m. to 12.25 p.m. everyday school life, 12.25 p.m. lunch with a high GI-rice or a low GI-rice and a water beverage, 12.45 p.m. to 13.15 p.m. regular lunch break, 13.15 p.m. computerized tests of executive cognitive and basal (alertness) functioning.

Parameters of cognition with relevance to everyday school life are measured by a computerized test program developed by the Institute of Working Learning and Aging (ALA). Usual eating behaviour, sleep behaviour, physical activity and parental education were determined as control variables by questionnaires for children, parents.

ELIGIBILITY:
Inclusion Criteria:

* all fifth and sixth grade students of Gesamtschule Berger Feld with the consent of parents and child

Exclusion Criteria:

* Metabolic diseases or special diet

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Shifting: Change of total reaction time for a) [ms] | participants were tested on two test days (T1 and T2) with one week wash out
  Measuring global task-switching costs by a three-part computer trial.
  a. Non-switch: digits from 1 to 26 in random order are to put in order. b. Non-switch: Same as a) with letters from A to Z c. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
Shifting: Change of total reaction time for b) [ms | participants were tested on two test days (T1 and T2) with one week wash out
  Measuring global task-switching costs by a three-part computer trial.
  a. Non-switch: digits from 1 to 26 in random order are to put in order. b. Non-switch: Same as a) with letters from A to Z c. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
Shifting: Change of total switch-costs [ms | participants were tested on two test days (T1 and T2) with one week wash out
  Measuring global task-switching costs by a three-part computer trial.
  a. Non-switch: digits from 1 to 26 in random order are to put in order. b. Non-switch: Same as a) with letters from A to Z c. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
updating: change of ratio of missing [%] | participants were tested on two test days (T1 and T2) with one week wash out
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
updating: change of ratio of false alarms [%] | participants were tested on two test days (T1 and T2) with one week wash out
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
updating: change of mean reaction time [ms] | participants were tested on two test days (T1 and T2) with one week wash out
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
tonic alertness: change of mean reaction time [ms] | participants were tested on two test days (T1 and T2) with one week wash out
  measures the level of alertness in response to a simple visual stimulus. Mean reaction time
tonic alertness: change of deviation of reaction time [ms] | participants were tested on two test days (T1 and T2) with one week wash out
  measures the level of alertness in response to a simple visual stimulus. Deviation of reaction time
tonic alertness:change of numbers of omission errors [n] | participants were tested on two test days (T1 and T2) with one week wash out
  measures the level of alertness in response to a simple visual stimulus. subsidiary outcome is the numbers of omission errors.
tonic alertness:change of numbers of commission errors [n] | participants were tested on two test days (T1 and T2) with one week wash out
  measures the level of alertness in response to a simple visual stimulus. subsidiary outcome is the numbers of comission errors.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kersting, Prof, Study Chair — Research Institut of Child Nutrition
Locations (1):
- Germany Research Institute of Child Nutrition, Dortmund, Dortmund, Germany

IPD SHARING:
Plan to Share IPD: No